CLINICAL TRIAL: NCT06424028
Title: Presentation, Management, Hospital-course, and Prognosis of Acute Right Ventricular Infarction: A Prospective Registry of Patients Presenting to the Largest Primary Percutaneous Coronary Intervention Centre of Pakistan
Brief Title: Acute Right Ventricular Infarction Registry
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Rajesh Kumar, Associate Professor Adult Cardiology, National Institute of Cardiovascular Diseases, Pakistan
Other Study IDs: IRB-62/2023
Record Dates: First submitted 2024-05-10; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Inferior Wall; Transmural Myocardial Infarction; Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Right Ventricular Infarct — Consecutive patients presented with isolated inferior, infero-posterior and inferolateral wall MI with or without acute right ventricular infarction.

SUMMARY:
This Study aims to provide an assessment of clinical presentation, management, hospital course, and prognosis of acute right ventricular infarction presenting with or without Inferior or infero-posterior wall Myocardial Infarction and the assessment of composite adverse clinical outcome after reperfusion in-hospital and post-discharge (in 30 Days Prognosis).

DETAILED DESCRIPTION:
After fulfilling the eligibility criteria, informed consent will be obtained from all the patients regarding using data for research while maintaining anonymity.Data will be collected for various patient, system, and procedure related characteristics with the help of a predefined structured proforma consisted of demographic data, clinical presentation, history and co-morbid conditions, and angiographic and procedural characteristics. All the recruited patients will be kept under observiton during the hospital stay and a telephonic follow-up will be carried out after 30-days of discharge and occurrence of the MACE will be recorded.

Univariate and multivariable binary logistic regression analysis will be performed to determine the clinical predictors of RVI. Odds ratio (OR) along with 95% confidence interval (CI) will be reported. The statistical significance criteria will be set as p-value<0.05.

For data verification, 10% of the data will be cross-checked with the source document (Patient file).

ELIGIBILITY:
Inclusion Criteria:

* Patients of Inferior, infero-lateral and infero-posterior wall MI with and without RV infarction undergoing PPCI.
* Both male and female patients.
* Patients of age ≥ 18 years.

Exclusion Criteria:

• Patients who will not give consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented at a tertiary care hospital with Inferior and posterior wall MI with and without RV infarction undergoing PPCI who are fulfilling the eligibility criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-07-19 (Estimated); Study Completion 2024-08-19 (Estimated)

PRIMARY OUTCOMES:
Composite adverse clinical outcome | Upto 30 days from admission
  Atleast one adverse event, such as pump failure, cerebrovascular accident (CVA), stent thrombosis, major bleeding, contrast-induced nephropathy (CIN), ventricular arrhythmias, or mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Kumar, MBBS, FCPS, Principal Investigator — National Institute of Cardiovascular Diaseses
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The Hospital Medical Record number will be used as the patient identifier.